CLINICAL TRIAL: NCT02923752
Title: Whole Brain Vessel Wall Imaging in Stroke Patients (WISP): An International Multi-Center Registry
Acronym: WISP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Zhaoyang Fan, PhD, Technical Director, 3T MRI, Biomedical Imaging Research Institute, Cedars-Sinai Medical Center
Other Study IDs: 46315
Record Dates: First submitted 2016-10-03; First posted 2016-10-05 (Estimated); Last update posted 2018-08-14 (Actual); Status verified 2018-08

CONDITIONS: Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: Yes

INTERVENTIONS:
Device: MRI — Contrast-enhanced MRI

SUMMARY:
This is a new vessel wall imaging-based stroke registry which will investigate the clinical utility of the whole-brain intracranial vessel wall Magnetic Resonance Imaging (MRI) technique in assessing the etiologies in patients with ischemic stroke.

DETAILED DESCRIPTION:
The registry will focus on investigating the utility of whole-brain vessel wall MRI techniques in assessing the etiologies in patients with recent ischemic stroke. Patients who have had ischemic stroke (as confirmed by diffusion weighted MRI) and have had or will undergo 3D whole-brain vessel wall MRI within 8 weeks of symptom onset will be recruited into this study. It is anticipated that a total of 1000 subjects will be recruited from Feb 2017 to Feb 2019. Approximately 12 centers in the US and China will participate in the registry. MRI whole-brain vessel wall images will be analyzed for detection and characteristics of various vessel wall pathologies and association between vessel wall imaging findings and patient's clinical information.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥ 18 years of age
* Ischemic stroke onset within 8 weeks and confirmed by diffusion weighted MRI
* Ability to read and understand informed consent

Exclusion Criteria:

* The cause of stroke has been confirmed to be related to cardiac or extracranial carotid or aorta pathologies.
* Contraindications to MR imaging including mechanically, magnetically, or electrically activated implants, ferromagnetic implants and ferromagnetic foreign bodies, pregnancy.
* Inability to tolerate MRI imaging secondary to an inability to lie supine or severe claustrophobia.
* Non-compliant with visit instructions, including inability to lie still, hold breath or follow procedure instructions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients had recent ischemic stroke and have had or will undergo 3D whole-brain vessel wall MRI within 8 weeks of symptom onset.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2017-02-01 (Actual); Primary Completion 2019-08-01 (Estimated); Study Completion 2019-08-01 (Estimated)

PRIMARY OUTCOMES:
Vessel wall pathology findings by MRI | baseline
  To identify vessel wall pathologies such as atherosclerosis, dissection, vasculitis

CONTACTS AND LOCATIONS:
Overall Officials: Zhaoyang Fan, PhD, Principal Investigator — Cedars-Sinai Medical Center; Qi Yang, MD,PhD, Principal Investigator — Cedars-Sinai Medical Center; Debiao Li, PhD, Principal Investigator — Cedars-Sinai Medical Center
Locations (12):
- United States (3):
  - Keck Hospital of the University of Southern California, Los Angeles, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Torrance Memorial Medical Center, Torrance, California
- China (9):
  - LiangXiang Hospital, Beijiang
  - Chaoyang Hospital, Capital Medical University, Beijing
  - Beijing AeroSpace Center Hospital, Beijing
  - Xuanwu Hospital, Capital Medical University, Beijing
  - West China Hospital, Sichuan University, Chengdu
  - Fujian Medical University Union Hospital, Fuzhou
  - Tianjin First Center Hospital, Tianjin
  - Tianjin Huanhu Hospital, Tianjin
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Fan Z, Yang Q, Deng Z, Li Y, Bi X, Song S, Li D. Whole-brain intracranial vessel wall imaging at 3 Tesla using cerebrospinal fluid-attenuated T1-weighted 3D turbo spin echo. Magn Reson Med. 2017 Mar;77(3):1142-1150. doi: 10.1002/mrm.26201. Epub 2016 Feb 28. PMID 26923198
- [Result] Bodle JD, Feldmann E, Swartz RH, Rumboldt Z, Brown T, Turan TN. High-resolution magnetic resonance imaging: an emerging tool for evaluating intracranial arterial disease. Stroke. 2013 Jan;44(1):287-92. doi: 10.1161/STROKEAHA.112.664680. Epub 2012 Nov 29. No abstract available. PMID 23204050